CLINICAL TRIAL: NCT07348913
Title: Impact of Regular Low-Frequency Hemoperfusion on Medium- to Long-Term Prognosis in Maintenance Dialysis Patients: A Real-World Single-Center Retrospective Study
Brief Title: Impact of Regular Low-Frequency Hemoperfusion on Medium- to Long-Term Prognosis in Maintenance Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Yunfeng Xia (Other)
Responsible Party: Sponsor-Investigator, Yunfeng Xia, Chief Physician of Nephrology、Clinical Professor, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: Chong qing Medical University
Record Dates: First submitted 2025-12-29; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-01

CONDITIONS: Regular Low-Frequency Hemoperfusion; Medium- to Long-Term Prognosis; Maintenance Dialysis Patients; Retrospective Study
Keywords: Hemoperfusion; Maintenance Dialysis; Propensity Score Matching; Survival Analysis; Competing Risk; Cardiovascular/Cerebrovascular Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hemoperfusion group: receive regular low-frequency hemoperfusion once monthly
- non-hemoperfusion group: not receive regular low-frequency hemoperfusion once monthly

SUMMARY:
Objective: To investigate the effect of regular low-frequency hemoperfusion on all-cause mortality and cardiovascular/cerebrovascular mortality risk in maintenance hemodialysis (MHD) patients.

Methods: Data from MHD patients over the past 10 years at our blood purification center were retrospectively collected. Patients were divided into a hemoperfusion group (receiving regular low-frequency hemoperfusion once monthly) and a non-hemoperfusion group. Propensity score matching (PSM) was used to balance baseline characteristics. Differences in cumulative all-cause and cardiovascular/cerebrovascular mortality between the two groups before and after matching were compared. A competing risk model was employed to analyze mortality risk.

DETAILED DESCRIPTION:
Clinical and laboratory data were collected for all enrolled patients. These included age, sex, underlying medical conditions, dialysis vintage, blood pressure, serum albumin, hemoglobin, platelet count, C-reactive protein (CRP), serum calcium, serum phosphorus, intact parathyroid hormone (iPTH), total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), triglycerides, and serum β2-microglobulin. Time-averaged mean values were calculated for blood pressure and laboratory parameters across the entire follow-up period. Data on cardiovascular/cerebrovascular death and all-cause mortality over the past ten years were also compiled.

Given the considerably larger size of the Hemoperfusion Group compared with the Non-Hemoperfusion Group, propensity score matching (PSM) was performed by specialized statisticians during data processing to balance baseline characteristics between the two groups. This approach enabled a systematic assessment of the effect of regular low-frequency hemoperfusion on cardiovascular/cerebrovascular and all-cause mortality in MHD patients.

ELIGIBILITY:
Inclusion criteria:

* Included patients were aged ≥18 years
* Undergo dialysis treatment three times a week (each session lasting 3-4 hours)
* Having basically complete clinical and laboratory records, and having received at least 6 months of follow-up at this center

Exclusion Criteria:

* Under 18 years old
* Does not receive dialysis three times a week (each session lasts 3-4 hours)
* Does not have basic complete clinical and laboratory records, and has not been followed up at this center for at least 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received MHD treatment at the Hemodialysis Center of the First Affiliated Hospital of Chongqing Medical University from January 2015 to December 31, 2024. Included patients were aged ≥18 years, received dialysis three times a week (each session lasting 3-4 hours), had basically complete clinical and laboratory records, and were followed up at our center for at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 879 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiovascular/Cerebrovascular Death | 1, 3, 5, and 10 years
all-cause mortality | 1, 3, 5, and 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No